CLINICAL TRIAL: NCT06908109
Title: Continuous Oral Suctioning During Flexible Bronchoscopy: Effect on Sedative Medication Needs and Both Endoscopist's and Patient's Satisfaction
Brief Title: This Study Will Evaluate the Effectiveness of a Simple Intervention Through a Classical Yankauer Oral Suction Tube, in Decreasing the Sedative Medication Doses Needed to Provide Effective Patient Sedation During Bronchoscopy, Along With Its Effect on Both Patient's and Bronchoscopist Satisfaction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Principal Investigator, Rayan Mohamad, Clinical Associate, American University of Beirut Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: IM.IBA.03
Record Dates: First submitted 2025-03-21; First posted 2025-04-03 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Bronchoscopy
MeSH Terms: interventions — Bronchoscopy

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sham Group (Sham Comparator): The control group: included another 60 patients, who underwent the regular FB procedure with a blinded defective Yankauer suction device (Sham) attached to the oral cavity of the patient and present throughout the procedure.
  Interventions: Procedure: Bronchoscopy
- Yankauer group (Active Comparator): The intervention group: included 60 patients, who underwent the regular FB procedure with a functional standard Yankauer suction device attached to the oral cavity of the patient and present throughout all the procedure.
  Interventions: Device: Yankauer Suction Device; Procedure: Bronchoscopy

INTERVENTIONS:
Device: Yankauer Suction Device — The Yankauer suction device is a hollow, curved and flexible tube that has a suction tip surrounded by a bulbous head to allow effective suctioning without damaging the surrounding tissue. It has been frequently used in multiple settings that range from minor dental procedures to large surgeries. It is also frequently used in the intensive care units to suction oropharyngeal secretions and prevent aspiration. Throughout this study, and regardless of the study group (control or intervention group), the Yankauer suction device is attached to a distinct suction port and placed, at the other end, inside the oral cavity of the patient.
  Arms: Yankauer group
Procedure: Bronchoscopy — Flexible bronchoscopy done for the following indications: presence of a lung mass or collapse, persistent pulmonary infiltrates, pulmonary infection in the setting of immunosuppression, hemoptysis, or other rare causes like chronic cough. Flexible bronchoscopy (FB) is a medical procedure that has been used for more than five decades for the diagnostic evaluation and/or therapeutic intervention in a multitude of pulmonary and bronchial diseases

SUMMARY:
The aim of this study is to evaluate the effectiveness of a simple intervention through a classical Yankauer oral suction tube, a device known to have a proven safety profile in multiple healthcare settings, in decreasing the sedative and opioid medication doses needed to provide effective patient sedation during bronchoscopy, along with its effect on both patient's and bronchscopist's satisfaction throughout the procedure.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or above
* inpatients or outpatients
* scheduled to have a flexible bronchoscopy for one of multiple indications based on their physician's assessment, including the presence of a lung mass or collapse, persistent pulmonary infiltrates, pulmonary infection in the setting of immunosuppression, hemoptysis, or other rare causes like chronic cough.
* patients provided a written informed consent.

Exclusion Criteria:

* patients with anatomic oro-pharyngeal abnormalities,
* critically ill patients
* uncooperative patients or inability to provide signed consent by the patient or their legal representative
* coagulopathy or bleeding diathesis
* severe obstructive airway disease
* recent myocardial infarction
* uncontrolled or poorly controlled asthma or chronic obstructive pulmonary disease (COPD)
* pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2016-03-04 (Actual); Primary Completion 2022-10-14 (Actual); Study Completion 2022-10-14 (Actual)

PRIMARY OUTCOMES:
Mean doses of Midazolam and Fentanyl | From enrollment (pre-bronchoscopy) to the end of the bronchoscopic procedure (up to 30 minutes)
  From the time of enrollment (pre-bronchoscopy) to the end of the bronchoscopic procedure

IPD SHARING:
Plan to Share IPD: No